CLINICAL TRIAL: NCT04310566
Title: Evaluation of a Daily Disposable Novel Multifocal Contact Lens in a Myopic Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6385
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Results first posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2021-12

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Test/Control (Experimental): Eligible subjects that are habitual soft contact lenses will be randomized into one of the two possible lens wear sequences: Test/Control or Control/Test
  Interventions: Device: JJVC Investigational Multifocal Contact Lens (senofilcon A c3); Device: Dailies Total 1® Multifocal Contact Lens
- Control/Test (Experimental): Eligible subjects that are habitual soft contact lenses will be randomized into one of the two possible lens wear sequences: Test/Control or Control/Test
  Interventions: Device: JJVC Investigational Multifocal Contact Lens (senofilcon A c3); Device: Dailies Total 1® Multifocal Contact Lens

INTERVENTIONS:
Device: JJVC Investigational Multifocal Contact Lens (senofilcon A c3) — TEST
Device: Dailies Total 1® Multifocal Contact Lens — CONTROL

SUMMARY:
This is a single-masked, crossover, randomized-controlled, dispensing clinical trial. A total of approximately 70 myopic eligible subjects will be targeted to complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study.

  1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. The subject must be at least 40 years of age and not greater than 70 years of age at the time of consent.
  4. Subjects must own a wearable pair of spectacles if required for their distance vision.
  5. The subject must be an adapted soft contact lens wearer in both eyes (i.e. worn lenses a minimum of 2 days per week for at least 6 hours per wear day, for 1 month or more duration).
  6. The subject must either already be wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or, if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire".
  7. The subject's distance spherical equivalent refraction must be in the range of -1.25 D to -3.75 D in each eye.
  8. The subject's refractive cylinder must be ≤0.75 D in each eye.
  9. The subject's ADD power must be in the range of +0.75 D to +2.50 D.
  10. The subject must have distance best corrected visual acuity of 20/20-3 or better in each eye.

      Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or lactating.
  2. Any active or ongoing ocular or systemic allergies that may interfere with contact lens wear.
  3. Any active or ongoing systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
  4. Any previous, or planned, ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, lid procedures, cataract surgery, retinal surgery, etc.).
  5. A history of amblyopia, strabismus or binocular vision abnormality.
  6. Use of any of the following oral medications within 2 weeks prior to enrollment: oral retinoids, oral tetracyclines, anticholinergics, systemic/topical steroids. See section 9.1 for additional details regarding excluded systemic medications.
  7. Use of any ocular medication, with the exception of rewetting drops.
  8. History of herpetic keratitis.
  9. History of irregular cornea.
  10. History of pathological dry eye.
  11. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
  12. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
  13. Any known hypersensitivity or allergic reaction to non-preserved rewetting drop solutions or sodium fluorescein.
  14. Clinically significant (Grade 2 or greater) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear.
  15. Entropion, ectropion, extrusions, chalazia, recurrent styes, dry eye, glaucoma, history of recurrent corneal erosions.
  16. Any current ocular infection or inflammation.
  17. Any current ocular abnormality that may interfere with contact lens wear.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2020-03-28 (Actual); Study Completion 2020-03-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Dr. James Weber & Associates, PA, Jacksonville, Florida
  - VRC-East, Jacksonville, Florida
  - Maitland Vision Center, Maitland, Florida
  - Kannarr Eye Care, Pittsburg, Florida
  - Visual Eyes, Roswell, Georgia
  - ProCare Vision Centers, Granville, Ohio
  - West Bay Eye Associates, Warwick, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 67 subjects were enrolled into this study. Of those enrolled, 65 were dispensed at least one study lens, while 2 subjects failed to meet all eligibility criteria. Of those dispensed a study lens, 17 subjects completed the study prior to the study being terminated, while 45 subjects were discontinued. This study was terminated due to the COVID-19 Pandemic.
Groups:
- Test/Control: Subjects randomized to this sequence received the Test lens during the first period and then received the Control lens during the second period
- Control/Test: Subjects randomized to this sequence received the Control lens during the first period and then received the Test lens during the second period
Period: Period 1
Arm/Group | Test/Control | Control/Test
Started | 31 | 34
Completed | 15 | 14
Not Completed | 16 | 20
Not completed — Study Termination due to COVID-19 | 15 | 17
Not completed — Protocol Violation | 0 | 1
Not completed — Subject no longer meets eligbility criteria | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Period: Period 2
Arm/Group | Test/Control | Control/Test
Started | 15 | 14
Completed | 8 | 9
Not Completed | 7 | 5
Not completed — Study Termination | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- All Dispensed Subjects: All subjects dispensed a study lens.
Arm/Group | All Dispensed Subjects
Number analyzed (Participants) | 65
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.3 (6.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  Black or African American | 8
  White | 56
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 65

OUTCOME MEASURES:

1. Primary Outcome: Subjective Vision Scores
Description: Subjective Overall Quality of Vision was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient- xperience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: 1-Week Follow-up
Population: All available data
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Test: All subjects that wore the Test lens during either the first or second period fo the study
- Control: All subjects that wore the Control lens during either the first or second period of the study.
Arm/Group | Test | Control
Number analyzed (Participants) | 28 | 31
Units on a Scale | 61.41 (19.917) | 55.03 (18.199)

2. Primary Outcome: Visual Acuity (logMAR)
Description: High contrast bright illumination binocular logMAR (Logarithm of the Minimum Angle of Resolution) visual acuity was assessed at distance (4 meters) using ETDRS Charts, near (40 cm) and intermediate (64 cm) using reduced Guillon-Poling charts. A value of 0.0 logMAR indicated a Snellen vision of 20/20. Lower logMAR visual acuity values indicates better vision. The average logMAR visual acuity for each lens was reported. Note: The room illuminance was required to be between 7.3 and 7.9 EV (394-597 lux). Acceptable Luminance Range for Distance (4M): 10.5-10.7 EV (181-208 cd/m2). Acceptable Luminance Range for Near (40cm) and Intermediate Guillon-Poling :10.8- 11.1 EV (223-274 cd/m2).
Time Frame: 1-Week Follow-up
Population: All avaiable data.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Test | Control
Number analyzed (Participants) | 28 | 31
logMAR
  Distance (4 meters) | -0.11 (0.116) | -0.11 (0.112)
  Intermediate (64 centimeters) | -0.09 (0.092) | -0.06 (0.093)
  Near ( 40 centimeters) | 0.01 (0.135) | 0.05 (0.129)

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study. Up to 2-Week Follow-up for subjects that completed study. Thirty-two subjects were monitored up to the 1-Week evaluation since the study was terminated early due to COVID-19.
Groups:
- Test: All subjects that wore the Test lens during either the first or second period of the study.
Arm/Group | Test | Control
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/49
Other Adverse Events (participants affected / at risk) | 0/45 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-05): https://cdn.clinicaltrials.gov/large-docs/66/NCT04310566/Prot_SAP_000.pdf